CLINICAL TRIAL: NCT07236229
Title: The Effects of Immersive Virtual Reality-Based Exercise Therapy on Pain, Functionality, Sleep, and Cognitive Functions in Patients With Grade 1-2 Adhesive Capsulitis
Brief Title: The Effects of Immersive Virtual Reality in Patients With Grade 1-2 Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Hande Besna Göçen, Lecturer, MSc Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BahcesehirU_H_AC-VR_01
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Adhesive Capsulitis; Virtual Reality; Sleep; Pain; Cognition
Keywords: Adhesive Capsulitis; Virtual Reality; Sleep; Pain; Cognition
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups using the stratified randomization method. The first group will be the immersive virtual reality-based exercise group (n=18), and the second group will be the conventional exercise group (n=18).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality-Based Exercise Therapy (Experimental): Participants in this group will receive immersive virtual reality-based exercise therapy using Oculus Quest 2 applications (Guided Tai Chi and Reach Shoulder Health) for 6 weeks, 2 sessions per week.
  Interventions: Other: Immersive Virtual Reality-Based Exercise Therapy
- Conventional Physiotherapy Group (Active Comparator): Participants in this group will receive standard physiotherapy exercises for adhesive capsulitis including ROM, stretching, and strengthening for 6 weeks, 2 sessions per week.
  Interventions: Other: Conventional Physiotherapy Group

INTERVENTIONS:
Other: Conventional Physiotherapy Group — In the conventional exercise group, participants will perform range of motion exercises, pendulum exercises, finger ladder exercises, stretching, and strengthening exercises. The traditional exercise therapy will be administered twice a week for six weeks, with each session lasting 30 minutes.
  In addition, both groups will receive identical patient education and home exercise programs. Patient education will be delivered face-to-face for 30 minutes at the beginning of the intervention. The home exercise program will be performed progressively at home on non-intervention days, five days per week.
  Arms: Conventional Physiotherapy Group
Other: Immersive Virtual Reality-Based Exercise Therapy — Patients in the immersive virtual reality-based exercise group will participate in the exercise program using the Oculus Quest 2 device. Sessions will be conducted twice a week for six weeks, each lasting 30 minutes. Two different virtual reality applications, Reach Shoulder Health and Guided Tai Chi, will be administered to the patients in this group.
  In addition, both groups will receive identical patient education and home exercise programs. Patient education will be delivered face-to-face for 30 minutes at the beginning of the intervention. The home exercise program will be performed progressively at home on non-intervention days, five days per week.
  Arms: Immersive Virtual Reality-Based Exercise Therapy

SUMMARY:
Adhesive capsulitis (frozen shoulder) is a complex condition characterized by inflammation, fibrosis, and restriction of movement in the shoulder capsule, significantly limiting an individual's participation in daily living activities. It is most commonly observed in individuals aged between 40 and 60 years, and its treatment frequently involves approaches such as manual therapy, exercise, corticosteroid injections, and electrotherapy. However, these conventional methods may be limited by factors such as lack of motivation, pain-related avoidance behavior, and poor treatment adherence.

Today, immersive virtual reality technologies introduce a new dimension to rehabilitation by gamifying exercise, providing sensory feedback, and enabling graded exposure through mechanisms such as distraction and engagement. They also enhance motivation and compliance with exercise programs. Studies in the literature have reported that virtual reality-based exercise is an effective method for reducing pain levels in patients diagnosed with frozen shoulder.

However, only a limited number of studies have specifically examined the effects of immersive virtual reality in patients with adhesive capsulitis. To date, no study has investigated the impact of immersive virtual reality interventions on sleep and cognitive functions in these patients. Furthermore, the combined effect of patient education, home exercise programs, and immersive virtual reality therapy has not yet been explored. For these reasons, the present study aims to investigate the effects of immersive virtual reality-based exercise therapy on pain, functionality, sleep, and cognitive functions in patients with Grade 1-2 adhesive capsulitis.

DETAILED DESCRIPTION:
Our study was designed as a single-center, randomized, controlled, prospective trial aiming to compare the effectiveness of immersive virtual reality-based exercise therapy and conventional therapy in patients diagnosed with Grade 1-2 adhesive capsulitis.Patients who consent to participate will be randomly assigned to two groups:

Intervention Group (n = 15): Patient education + Home exercise program + Immersive virtual reality-based exercise therapy

Control Group (n = 15): Patient education + Home exercise program + Conventional exercise therapy

Intervention Process All participants will receive treatment twice a week for six weeks, with each session lasting 30 minutes. The initial assessment will be conducted before the first session, and the final assessment will take place at the end of the sixth week. Both the immersive virtual reality-based exercise group and the conventional exercise group will receive patient education. The educational content aims to describe the natural course of the disease, promote activity modification to encourage functional and pain-free range of motion, and adjust stretching intensity to suit the patient's current level.

Patient education will be delivered once, face-to-face, for 30 minutes before the interventions begin, and it will cover five main topics:

Introduction to the Disease: General information about adhesive capsulitis. Pain Mechanisms and Perception: Education on pain pathways and interpretation. Encouragement of Activity: Emphasis on safely using the shoulder within pain-free limits during daily life activities.

Preparation for Treatment: Explanation that the virtual reality-based therapy will be conducted in a gamified and motivating environment, while the control group will receive traditional physiotherapy methods.

Exercise Adherence and Follow-up: Emphasis on the importance of active participation for treatment success and the monitoring of progress through pre- and post-assessments.

Hanchard et al. strongly supported the implementation of patient education and home exercise programs in individuals with adhesive capsulitis.

Home Exercise Program In addition to patient education, both groups will perform the same home exercise program. Participants will carry out the exercises at home for 30 minutes a day, five days a week, over a six-week period (on non-intervention days). The home exercise program will be progressive and similar to the conventional therapy applied by the physiotherapist. It will include range of motion (ROM) exercises, stretching exercises, and pendulum exercises.

Immersive Virtual Reality-Based Exercise Group In the immersive virtual reality group, the Oculus Quest 2 headset will be used with the Guided Tai Chi and Reach Shoulder Health applications, both applied progressively. Oculus Quest 2 is a virtual reality headset used for therapeutic purposes in shoulder rehabilitation and has been previously applied in patients with adhesive capsulitis.

The Template for Intervention Description and Replication (TIDieR) checklist and guide were used to describe the intervention protocols in detail, ensuring reproducibility and clinical applicability. Both the immersive virtual reality and conventional exercise intervention programs were developed in accordance with TIDieR recommendations.

The Reach Shoulder Health program is an interactive virtual reality application that gamifies shoulder rehabilitation exercises. It includes a variety of modules designed to enhance upper extremity range of motion, coordination, and muscle activation-particularly beneficial for patients with restricted shoulder mobility such as adhesive capsulitis. The program progressively trains shoulder mobilization, target-reaching, hand-eye coordination, range of motion, and muscle strengthening around the shoulder. Its game modules, including Firefly Assessment, Space Gunner, Bullseye, Tube Trouble, Star Beams, and Power Pop, are structured to be both entertaining and therapeutic, incorporating multiple levels to increase patient motivation and treatment adherence. Participants will progress through five levels each week over the six-week period.

The Guided Tai Chi application is another virtual reality program designed to enhance shoulder mobility and provide pain-free movement experiences while reducing anxiety and improving motivation in patients with adhesive capsulitis. The exercises in this application will also be progressively increased in difficulty across beginner, intermediate, and advanced levels throughout the six-week intervention.

Conventional Exercise Group Participants in the conventional exercise group will receive a 30-minute exercise session twice a week for six weeks. The program will include range of motion exercises, pendulum exercises, finger ladder activities, stretching, and strengthening exercises. All exercises will be applied progressively, increasing in intensity over time.

Evaluation All participants will be assessed for pain levels, shoulder range of motion, ability to perform daily living activities, sleep quality, and cognitive functions using valid and reliable measurement tools before and after the interventions. Assessments will be conducted at the first session and at the end of the sixth week, and pre- and post-intervention results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adhesive capsulitis by a doctor
* Classified as Grade 1-2 adhesive capsulitis
* Receiving physiotherapy for adhesive capsulitis for the first time
* Aged between 18 and 64 years
* Suitable for using a VR headset

Exclusion Criteria:

* Previous history of physiotherapy
* Presence of any mental disorder
* Recent surgery or any shoulder condition (e.g., fractures around the shoulder region) that contraindicates shoulder mobilization
* History of receiving injections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by the Visual Analog Scale (VAS) | Baseline and at the end of the 6-week intervention period
  The VAS assesses perceived shoulder pain intensity on a 10-cm line from "no pain" to "worst pain imaginable.

SECONDARY OUTCOMES:
Shoulder Function (Shoulder Pain and Disability Index - SPADI) | Baseline and at the end of the 6-week intervention period
  Shoulder pain and disability will be assessed with the SPADI, which evaluates pain and functional limitation on a 0-100 scale, where higher scores indicate greater impairment.
Shoulder Range of Motion (ROM) | Baseline and at the end of the 6-week intervention period
  Shoulder joint mobility (flexion, extension, abduction, adduction, internal and external rotation) will be measured in degrees using a goniometer to evaluate changes in movement capacity.
Pain Catastrophizing (Pain Catastrophizing Scale - PCS) | Baseline and at the end of the 6-week intervention period
  Catastrophic thinking related to pain will be assessed using the PCS, which measures rumination, magnification, and helplessness. Total scores range from 0 to 52, with higher scores indicating greater levels of pain catastrophizing.
Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | Baseline and at the end of the 6-week intervention period
  The PSQI assesses sleep quality over the past month across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Component scores (0-3) are summed to yield a global score (0-21), with higher scores indicating poorer sleep quality (commonly, >5 suggests poor sleep).
Digit Span Test | Baseline and at the end of the 6-week intervention period
  The Digit Span Test (DST) will be used to assess attention, short-term memory, and processing speed. It consists of two parts: Digit Span Forward (DSF) and Digit Span Backward (DSB). The total score ranges from 0 to 17 (maximum DSF = 9, DSB = 8). Higher scores indicate better verbal attention and short-term memory performance.
Wisconsin Card Sorting Test | Baseline and at the end of the 6-week intervention period
  Wisconsin Card Sorting Test (WCST) will be used to assess executive functions, including cognitive flexibility, abstract reasoning, and problem-solving ability. The primary outcome measures will include total errors, perseverative errors, and non-perseverative errors. Scores range from 0 to 128, with fewer errors indicating better executive functioning.
Benton Visual Retention Test | Baseline and at the end of the 6-week intervention period
  Benton Visual Retention Test (BVRT) will be used to assess short-term visual memory, visual perception, and visuoconstructive abilities. The version used in this study will be Form F, which will include 15 stimulus cards and 15 corresponding multiple-choice response cards.
  Scores will be calculated as the number of correct responses, with a possible range of 0 to 15. Higher scores will indicate better visual memory performance.
Virtual Reality Discomfort Questionnaire | At the end of the first Virtual Reality session
  Virtual Reality Discomfort Questionnaire includes symptoms such as fatigue, eyestrain, headache, and dizziness. Each item is rated on a 4-point Likert-type scale ranging from 0 (never) to 3 (very often). The total score is obtained by summing all item scores and then converting it into a percentage for interpretation. Higher scores indicate a greater level of discomfort associated with virtual reality use.
Virtual Reality Satisfaction Questionnaire | At the end of the first Virtual Reality session
  Virtual Reality Satisfaction Questionnaire will be used to provide descriptive data to understand the contribution of the virtual reality experience to the therapeutic process and patient comfort. The questionnaire consists of a total of 10 items under four subdimensions: ease of use, visual/auditory experience, engagement/interest, and overall satisfaction. Each item will be rated on a 4-point Likert-type scale ranging from 0 (never) to 3 (very often). The total score will be obtained by summing all item scores and converting the result into a percentage for interpretation. Higher scores will indicate greater patient satisfaction with the virtual reality experience.

CONTACTS AND LOCATIONS:
Overall Officials: Hande B Gocen, PhD (c), Principal Investigator — Istanbul Gelisim University
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing individual raw data is not appropriate due to ethical committee approval requirements and personal data protection regulations.

REFERENCES:
- [Background] Mena-Del Horno S, Balasch-Bernat M, Louw A, Luque-Suarez A, Rodriguez-Brazzarola P, Navarro-Ledesma S, Murillo C, Duenas L, Lluch E. Is there any benefit of adding a central nervous system-focused intervention to a manual therapy and home stretching program for people with frozen shoulder? A randomized controlled trial. J Shoulder Elbow Surg. 2023 Jul;32(7):1401-1411. doi: 10.1016/j.jse.2023.02.134. Epub 2023 Mar 29. PMID 37001795
- [Background] Mertens MG, Meert L, Struyf F, Schwank A, Meeus M. Exercise Therapy Is Effective for Improvement in Range of Motion, Function, and Pain in Patients With Frozen Shoulder: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2022 May;103(5):998-1012.e14. doi: 10.1016/j.apmr.2021.07.806. Epub 2021 Aug 21. PMID 34425089
- [Background] Hanchard NCA, Goodchild L, Brealey SD, Lamb SE, Rangan A. Physiotherapy for primary frozen shoulder in secondary care: Developing and implementing stand-alone and post operative protocols for UK FROST and inferences for wider practice. Physiotherapy. 2020 Jun;107:150-160. doi: 10.1016/j.physio.2019.07.004. Epub 2019 Jul 19. PMID 32026815
- [Background] Demir OB, Kablanoglu S, Sari PN, Alyanak B, Taskin Yilmaz F, Dursun E. Effects of virtual reality exercise on pain, joint motion, and quality of life in patients with frozen shoulder: a randomized controlled study. Physiother Theory Pract. 2025 Jul;41(7):1435-1446. doi: 10.1080/09593985.2024.2443027. Epub 2024 Dec 19. PMID 39700302
- [Background] Ozlu A, Ustundag S, Bulut Ozkaya D, Menekseoglu AK. Effect of Exergame on Pain, Function, and Quality of Life in Shoulder Impingement Syndrome: A Prospective Randomized Controlled Study. Games Health J. 2024 Apr;13(2):109-119. doi: 10.1089/g4h.2023.0108. Epub 2024 Feb 23. PMID 38394299